CLINICAL TRIAL: NCT02375061
Title: A Positive Psychology Intervention for Fibromyalgia Patients to Promote Physical and Psychological Wellbeing Using Information and Communication Technologies
Brief Title: A Positive Psychology Intervention for Fibromyalgia Patients Using ICT´s
Acronym: BPS_FM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UJaime011
Record Dates: First submitted 2015-02-16; First posted 2015-03-02 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-04

CONDITIONS: Fibromyalgia; Chronic Pain
Keywords: Best Possible Self; Positive Psychology; Optimism; Positive Technologies; Future thinking; Pain Catastrophizing
MeSH Terms: conditions — Fibromyalgia; Chronic Pain | interventions — Activities of Daily Living

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- e-BPS intervention (Experimental): Participants are asked to write and imagine about a future in which they have reached all their goals in four different domains: personal, professional, social and health domain. They carry out the exercise in a Positive Technology System called the "Book of Life", which has shown efficacy in the enhancement of positive mood (Baños, Etchemendy, Farfallini, García-Palacios, Quero & Botella, 2014). This application looks like a personal diary, where participants can write all that they want and these essays are supported by multimedia content (pictures, songs and videos). Additionally, they can continue doing the exercise in a web platform (TEO-Emotional Therapy Online) in which they can visualize all the content they had developed previously.
  Interventions: Behavioral: e-BPS
- Daily Activities (Placebo Comparator): Participants are asked to think and write about all that they have done the last 24 hours. They carry out the exercise in a powerpoint document, where they can record all the activities, situations and thoughts.
  Interventions: Behavioral: Daily Activities

INTERVENTIONS:
Behavioral: e-BPS
  Arms: e-BPS intervention
Behavioral: Daily Activities
  Arms: Daily Activities

SUMMARY:
This study is aimed to test the efficacy of a Positive Psychology Intervention (Best Possible Self, BPS) over optimism, future expectancies and positive affect at mid-term, in comparison to a control group, in fibromyalgia patients. The principal hypothesis is that the BPS intervention will enhance significantly the levels of optimism, positive future expectancies and positive affect in comparison to the Control group at short and mid-term.

DETAILED DESCRIPTION:
Previous studies have demonstrated the effects of positive psychological factors in pain adjustment. Specially, optimism has been linked to lower pain sensitivity, better physical functioning, less psychological distress and pain catastrophizing. Until recently, the beneficial effects of optimism on pain have been studied mostly in correlational studies or in experimental interventions in laboratory settings. To address the gap between research and clinical practice, the aim of this study is to test the efficacy of the Best Possible Self intervention (BPS) using Information and Communication Technologies (ICTs) with fibromyalgia patients.

BPS is a guided imagery exercise that requires participants to envision themselves in the future, achieving desired goals in different areas of their lives. This exercise has shown efficacy improving optimism, future expectancies and positive affect compared to a control condition, in general population (Meevissen, Peters & Alberts, 2011; Sheldon &Lyubomirsky, 2012; Peters, Flink, Boersma & Linton, 2010). Taking into account the prior literature, the aim of the present study is to carry out a randomized controlled study in order to replicate the findings about the effects of BPS on optimism, mood and affect in a chronic pain population. The exercise will be applied through a Positive Technology system and the effects will be analyzed during four months. The design employed in this study is similar to the used in other studies (Meevissen et al, 2011; Renner, Schwarz, Peters & Huibers, 2014; Sheldon & Lyubomirsky, 2006).

ELIGIBILITY:
Inclusion Criteria:

* Patients have to fulfill the American College of Rheumatology criteria for primary FMS.
* Sign a consent form stating their willingness to participate

Exclusion Criteria:

* Presence of another severe physical illness
* Presence of severe psychological disorders
* Be currently involved in another psychological treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory II | 4 months
  This is one of the most widely questionnaires used to evaluate severity of depression in pharmacological and psychotherapy trials. The instrument has good internal consistency (Cronbach's alpha of 0.76 to 0.95) and test-retest reliability of around 0.8. The Spanish version of this instrument has also shown a high internal consistency (Cronbach's alpha of 0.87) for both the general and the clinical population (Cronbach's alpha of 0.89). Summed to obtain the total score, which can be a maximum of 63 points.

SECONDARY OUTCOMES:
Pain Catastrophizing | 4 months
  The PCS instructions ask participants to reflect on past painful experiences, and to indicate the degree to which they experienced each of 13 thoughts or feelings when experiencing pain, on 5-point scales with the end points (0) not at all and (4) all the time. The PCS yields a total score and three subscale scores assessing rumination, magnification and helplessness. The PCS has been shown to have adequate to excellent 6 internal consistency (coefficient alphas: total PCS = 0.87, rumination = 0.87, magnification = 0.66, and helplessness = 0.78).
Positive and Negative Affect Scale | 4 months
  This measure analyzes the levels of positive (PA) and negative affect (NA). The instrument consists of 20 items, 10 for each level of affect. Participants rate on a 5-point scale (Not at all - Extremely). The Spanish version has demonstrated high internal consistency (0.89 to 0.91 for PA and NA in women and 0.87 for AP and 0.89 for AN in men) in college students.
Life Orientation Test | 4 months
  This scale measures positive and negative expectancies about future events. It consists of 20 statements referring to negative expectancies and 10 statements referring to positive expectancies. Participants answer on a 7-point scale (Not at all likely to occur - Extremely likely to occur). Some studies have found an appropriate levels of internal consistency for positive and negative expectancies (α=0.80-0.82 and 0.91, respectively).
Quality of Life | 4 months
  It consists of 10 items that evaluate perceived well-being in different areas (physical, psychological/emotional, occupational functioning, interpersonal functioning, among others)
Overall Anxiety Severity and Impairment Scale | 4 months
  OASIS is a brief instrument consisting of 5 items that measure the frequency and severity of anxiety, as well as the level of avoidance and work/school/home and social interference that anxiety produces.
General Self-Efficacy scale | 4 months
  This is a 12-item scale that evaluates perceived global self-efficacy and three main aspects of it: initiative, persistence and effort. All items are responded to on a 5-point scale, ranging from 1 (never happens to me) to 5 (always happens to me).
Subjective probability task | 4 months
  This scale measures positive and negative expectancies about future events. It consists of 20 statements referring to negative expectancies and 10 statements referring to positive expectancies. Participants answer on a 7-point scale (Not at all likely to occur - Extremely likely to occur). Some studies have found an appropriate levels of internal consistency for positive and negative expectancies (α=0.80-0.82 and 0.91, respectively).

OTHER OUTCOMES:
Fibromyalgia Impact Questionnaire | 4 months
  The FIQ-R is a 10-item self-report questionnaire that measures the health status of patients with FMS assessing the interference of FMS in their daily life.
Brief Symptom Inventory | Baseline
  It is a well validated self-report instrument for the measurement of general psychological distress.
Self concordance motivation | Baseline
  This questionnaire assess extrinsic and intrinsic motivation to practice the imagery exercise, rated on a 9-point scale ranging from 1 "not at all for this reason" to 9 "completely for this reason". SCM has been correlated withparticipants' frequency of practicing a daily imagery exercise and with self-reported imagery performance, a key aspect in self-applied interventions.
Eysenck Personality Questionnaire - Revised - Neuroticism | Baseline
  This scale assesses the neuroticism level of the individual, showing if he is stable or neurotic. This subscale is composed by 12 items of dicotomic response (yes-not). Regarding psychometric properties, studies found an alpha coefficient between 0.73 and 0.82.

CONTACTS AND LOCATIONS:
Overall Officials: Azucena García-Palacios, PhD, Principal Investigator — Universitat Jaume I
Locations (1):
- University Jaume I, Castellon, Castellón, Spain

REFERENCES:
- [Background] Meevissen YM, Peters ML, Alberts HJ. Become more optimistic by imagining a best possible self: effects of a two week intervention. J Behav Ther Exp Psychiatry. 2011 Sep;42(3):371-8. doi: 10.1016/j.jbtep.2011.02.012. Epub 2011 Mar 2. PMID 21450262
- [Background] Boselie JJLM, Vancleef LMG, Smeets T, Peters ML. Increasing optimism abolishes pain-induced impairments in executive task performance. Pain. 2014 Feb;155(2):334-340. doi: 10.1016/j.pain.2013.10.014. Epub 2013 Oct 19. PMID 24145210
- [Background] Hanssen MM, Vancleef LM, Vlaeyen JW, Peters ML. More optimism, less pain! The influence of generalized and pain-specific expectations on experienced cold-pressor pain. J Behav Med. 2014 Feb;37(1):47-58. doi: 10.1007/s10865-012-9463-8. Epub 2012 Oct 23. PMID 23239369
- [Background] Hanssen MM, Peters ML, Vlaeyen JWS, Meevissen YMC, Vancleef LMG. Optimism lowers pain: evidence of the causal status and underlying mechanisms. Pain. 2013 Jan;154(1):53-58. doi: 10.1016/j.pain.2012.08.006. Epub 2012 Oct 18. PMID 23084002
- [Background] Botella C, Riva G, Gaggioli A, Wiederhold BK, Alcaniz M, Banos RM. The present and future of positive technologies. Cyberpsychol Behav Soc Netw. 2012 Feb;15(2):78-84. doi: 10.1089/cyber.2011.0140. Epub 2011 Dec 9. PMID 22149078
- [Background] Sheldon, K. M., y Lyubomirsky, S. (2006). How to increase and sustain positive emotion: The effects of expressing gratitude and visualizing best possible selves. The Journal of Positive Psychology, 1(2), 73-82.
- [Background] Esteve-Vives J, Rivera Redondo J, Isabel Salvat Salvat M, de Gracia Blanco M, de Miquel CA. [Proposal for a consensus version of the Fibromyalgia Impact Questionnaire (FIQ) for the Spanish population]. Reumatol Clin. 2007 Jan;3(1):21-4. doi: 10.1016/S1699-258X(07)73594-5. Epub 2008 Nov 13. Spanish. PMID 21794391
- [Background] Garcia Campayo J, Rodero B, Alda M, Sobradiel N, Montero J, Moreno S. [Validation of the Spanish version of the Pain Catastrophizing Scale in fibromyalgia]. Med Clin (Barc). 2008 Oct 18;131(13):487-92. doi: 10.1157/13127277. Spanish. PMID 19007576
- [Background] MacLeod AK. Affect, emotional disorder, and future-directed thinking. Cognition & Emotion 10: 69-86, 1996.
- [Background] Mezzich JE, Ruiperez MA, Perez C, Yoon G, Liu J, Mahmud S. The Spanish version of the quality of life index: presentation and validation. J Nerv Ment Dis. 2000 May;188(5):301-5. doi: 10.1097/00005053-200005000-00008. PMID 10830568
- [Background] Bentley KH, Gallagher MW, Carl JR, Barlow DH. Development and validation of the Overall Depression Severity and Impairment Scale. Psychol Assess. 2014 Sep;26(3):815-830. doi: 10.1037/a0036216. Epub 2014 Apr 7. PMID 24708078
- [Background] Peters ML, Flink IK, Boersma K, Linton SJ. Manipulating optimism: can imagining a best possible self be used to increase positive future expectancies? Journal of Positive Psychology 5: 204-211, 2010.
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Scheier MF, Carver CS, Bridges MW. Distinguishing optimism from neuroticism (and trait anxiety, self-mastery, and self-esteem): a reevaluation of the Life Orientation Test. J Pers Soc Psychol. 1994 Dec;67(6):1063-78. doi: 10.1037//0022-3514.67.6.1063. PMID 7815302